CLINICAL TRIAL: NCT06144788
Title: A Randomized, Double-blind, Placebo-controlled, Parallel-group, Multicenter, Therapeutic Exploratory Phase 2 Study to Evaluate the Efficacy and Safety of JP-2266 in Patients With Type 2 Diabetes Mellitus
Brief Title: Evaluation of Efficacy and Safety When Administered JP-2266 in Type 2 Diabetes Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Jeil Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: JP-2266-201
Record Dates: First submitted 2023-11-13; First posted 2023-11-22 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Sodium-Glucose Transporter 2 Inhibitors

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- JP-2266 Low-dose (Experimental): Subjects take the investigational products once a day for 12 weeks.
  Interventions: Drug: SGLT2 inhibitor
- JP-2266 High-dose (Experimental): Subjects take the investigational products once a day for 12 weeks.
  Interventions: Drug: SGLT2 inhibitor
- placebo (Experimental): Subjects take the investigational products once a day for 12 weeks.
  Interventions: Drug: SGLT2 inhibitor

INTERVENTIONS:
Drug: SGLT2 inhibitor — SGLT 1/2 dual inhibitor
  Other Names: SGLT 1/2 dual inhibitor

SUMMARY:
A Randomized, Double-blind, Placebo-controlled, Parallel-group, Multicenter, Therapeutic Exploratory Phase 2 Study to Evaluate the Efficacy and Safety of JP-2266 in Patients with Type 2 Diabetes Mellitus

DETAILED DESCRIPTION:
Evaluation of efficacy and safety when administered JP-2266 in type 2 diabetes patients

ELIGIBILITY:
Inclusion Criteria:

1. Adult aged 19 to 80 years
2. Those diagnosed with type 2 diabetes
3. A person who provides diet and exercise therapy for the management of diabetes from 8 weeks before the screening criteria and can continue diet and exercise therapy during the clinical trial
4. Screening Results of the following criteria

   * 7% ≤ HbA1c ≤ 10%
   * FPG ≤ 270 mg/dL
5. Patients with 20 < BMI ≤ 45 kg/㎡
6. Those who voluntarily signed the informed consent to participate in this study

Exclusion Criteria:

1. Any type of diabetes other than type 2 diabetes
2. Screening when the inspection meets the following criteria

   * AST or ALT more than 3 times the normal upper limit
   * Total bilirubin exceeds twice the normal upper limit
   * eGFR < 60 mL/min/1.73㎡
3. A person with the following medical history or history of surgery/therapy

   * Medically significant history of kidney disease: kidney vascular obstruction disease, nephrectomy, kidney transplantation, etc
   * History of severe gastrointestinal surgery: total gastrectomy, total colon resection, small intestine resection, gastrointestinal anastomosis, gastrointestinal bypass, etc
   * history of acute pancreatitis or pancreatic surgery
   * History of undergoing bariatric surgery within 2 years before screening
   * Diabetic ketoacidosis, diabetic coma or whole marriage within 1 year prior to screening
   * Urinary tract infections or genital infections within 1 year prior to screening
   * Alcohol or drug addiction within 1 year prior to screening
   * A history of severe heart disease (heart failure, unstable angina, myocardial infarction, congestive heart failure symptoms
   * A person who has a history of significant surgery that causes electrolyte imbalance within 12 weeks before screening, or who is scheduled to undergo significant surgery within 12 weeks after the end of the clinical trial
   * Hypertension emergency medical history within 12 weeks prior to screening
   * There is a weight change of more than 10% within 12 weeks prior to screening, and symptoms of polyuria and bipolar disorder
   * A person with a history of malignancy within 5 years prior to screening However, a complete cure or properly controlled basal cell cancer, squamous cell skin cancer, or cervical intraepithelial cancer is allowed, but the history of bladder cancer cannot participate even if it has been more than 5 years
4. A person who has the following diseases or signs

   * Dysuria that is not medically controlled due to tense urinary incontinence, neurotic bladder, prostate hypertrophy, or symptoms of anuria, oliguria, urinary retention
   * Severe diabetic complications (proliferative diabetic retinopathy, nephropathy above stage 4 or severe diabetic neuropathy)
   * Chronic diseases that require continuous use of diuretics, systemic steroids or immunosuppressants (alveolar administration, injection)
   * Active liver disease, hepatitis, liver failure or cirrhosis
   * Patients with pituitary or adrenal insufficiency
   * Severe infections requiring the use of persistent antibiotics or immunotherapy drugs, and significant clinically trauma
   * an unstable mental illness that is not medically controlled
   * Severe gastrointestinal diseases: active ulcers, gastrointestinal/intestinal bleeding, active inflammatory bowel syndrome, patients with biliary obstruction, active gastritis not controlled by medication, etc
5. A person who has a history of hypersensitivity to the ingredients of a clinical trial drug, SGLT1/SGLT2 inhibitor or SGLT-2 inhibitor
6. Pregnant or lactating women
7. Participants in interventional clinical trials subject to other IP or medical devices within 12 weeks prior to screening
8. If the investigator is deemed unsuitable for the subject of this clinical trial due to other reasons

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Estimated)
Dates: Start 2023-11 (Estimated); Primary Completion 2024-03 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Changes in HbA1c at the 12 week from the baseline | 12 week

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Seoul, Seodaemun-gu, South Korea